CLINICAL TRIAL: NCT06217874
Title: Collection of Specimens and Clinical Data for Patients With Recurrent or Metastatic Breast Cancer or Male Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 14-002919; NCI-2023-10076 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14-002919 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2024-01-03; First posted 2024-01-23 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Breast Carcinoma; Metastatic Breast Carcinoma; Recurrent Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue specimens will be frozen and stored in the Biospecimen Accessioning and Processing Lab at Mayo Clinic Rochester. Part of the tissue specimen may be grown in the lab as organoids, which can be used to test drug responses, and some may be used to make xenografts-a process where part of the specimen is injected into mice to grow a new tumor used for future sequencing and drug studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo blood sample collection, provide clinical residual tissue samples and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being done to create a resource of samples and information that can be used to improve our understanding of the development, progression and treatment of recurrent or metastatic breast cancer or male breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To collect blood samples and fresh tissue from biopsies of metastatic lesions from Mayo Clinic patients with metastatic breast cancer.

OUTLINE: This is an observational study.

Patients undergo blood sample collection, provide clinical residual tissue samples and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Female participants must have histologically or cytologically confirmed invasive breast cancer.
* Male participants must have biopsy proven breast cancer.
* Age must be >= 18 years, and all must be able to understand and willing to sign an informed consent document.

Exclusion Criteria:

* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent; a history of serious or life-threatening allergic reaction to local anesthetics (i.e. lidocaine, xylocaine).
* Any other condition, which in the opinion of the patient's treating oncologist, or the physician performing the biopsy procedure, would make participation in this protocol unreasonably hazardous for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with invasive cancer, suspected or known recurrent or metastatic lesions, as well as males with biopsy proven breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-06-05 (Actual); Primary Completion 2034-06-30 (Estimated); Study Completion 2034-06-30 (Estimated)

PRIMARY OUTCOMES:
Response to targeted therapies | Baseline
  Response to targeted therapies will be evaluated in organoid or mouse xenograft models derived from tumor biospecimens obtained from participants.
Change in tumor cells | Baseline
  Changes in tumor cells will be evaluated following metastasis to other organs and after various treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Fergus J. Couch, Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials